CLINICAL TRIAL: NCT06640205
Title: Clinical and Radiographic Assessment of I-PRF Versus Nano Mineral Trioxide Aggregate Combined with I-PRF Scaffold in Vital Pulp Therapy in Mandibular First Molars with Closed Apices: "Randomized Controlled Trial"
Brief Title: Assessment of I-PRF Versus Nano MTA Combined with I-PRF Scaffold in Vital Pulp Therapy in Mature Mandibular First Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Elsayed Metwally Omar, Principle investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (32)/8-2023
Record Dates: First submitted 2024-08-16; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pulpotomy
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MTA Pulpotomy (Active Comparator): using MTA as pulpotomy capping agent in mature permanent teeth
  Interventions: Procedure: pulpotomy
- I-PRF pulpotomy (Experimental): using I-PRF as pulpotomy capping agent in mature permanent teeth
  Interventions: Procedure: pulpotomy
- I-PRF combined with Nano MTA pulpotomy (Experimental): using nano MTA mixed with I-prf as pulpotomy capping agent in mature permanent teeth
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: pulpotomy — Removal of coronal pulp tissue and then placing pulpotomy agent
  Other Names: full pulpotomy; vital pulp therapy

SUMMARY:
Assessment of I-PRF versus Nano Mineral trioxide aggregate Combined with I-PRF in pulpotomy in mature Mandibular First Molars

DETAILED DESCRIPTION:
Clinical and Radiographic Assessment of I-PRF versus Nano Mineral trioxide aggregate Combined with I-PRF Scaffold in Vital Pulp Therapy in Mandibular First Molars with Closed Apices: "Randomized Controlled Trial"

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Symptomatic irreversible pulpitis in mature mandibular molars only will be involved.

  * Patients of either gender aged from 15-30.
  * Tooth should give positive response to cold test.
  * The tooth is restorable
  * Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
  * Patients who will agree to the consent and will commit to follow-up period.
  * Patients with mature root.
  * Patients with no internal or external resorption and no periapical lesions.
  * Soft tissues around the tooth are normal with no swelling or sinus tract.

Exclusion Criteria:

* Patients with immature roots.

  * Haemostasias after 10 minutes can not be controlled after total pulpotomy
  * Patients with periapical lesions or infections.
  * Pregnant females.
  * Patients with fistula or swelling
  * Patients with necrotic pulp.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Post operative pain assessments | 6 hours post operative , 12 hours post operative , 24h (one day) post operative , 72h (3 days ) post operative and 7 days (one week) post operative
  Pain assessments were made postoperatively with numerical rate scale. The scale includes scores from 0 to 10 where 0 indicates no pain , scores 1 to 3 indicates mild pain , scores 4 to 6 indicates moderate and scores 7 to 10 indicates severe pain.

SECONDARY OUTCOMES:
Clinical and radiographic success | 1 month post operative ,3 months clinical and radiograph ,6 months clinical and radiograph ,9 months clinical and radiograph and 12 months clinical and radiograph.
  Clinically success : this includes that the tooth must be symptoms free ( No pain on percussion , no pain on biting and no pain with cold and hot ) . Also the tooth must not has any signs of failure as appearance of sinus tract or fistula during the follow up periods.
  Radiographic success : this includes that the tooth did not develop a periapical radiolucency as periapical periodontitis .
  Any deviation from the previous success criteria ( as clinical or radiographic ) considered as failure and the tooth will be shifted to root canal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Mo Omar, Master, Study Chair — Future University in Egypt
Locations (1):
- Future university in egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No